CLINICAL TRIAL: NCT01430819
Title: Safety and Immunogenicity Among Adults of Fluzone®, Influenza Virus Vaccine 2011-2012 Formulation (Intramuscular Route)
Brief Title: Study of Fluzone® Influenza Virus Vaccine 2011-2012 Formulation (Intramuscular Route) Among Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GRC48; U 1111-1120-1287 (Other: WHO)
Record Dates: First submitted 2011-09-07; First posted 2011-09-08 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2013-05

CONDITIONS: Influenza
Keywords: Influenza; Influenza Virus Vaccine; Fluzone® 2011-2012 Formulation; Fluzone® High-Dose 2011-2012 Formulation; Trivalent Inactivated Influenza Vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluzone® Vaccine Group (Experimental): Participants will receive the Influenza Virus Vaccine: Fluzone® 2011-2012 Formulation
  Interventions: Biological: Influenza Virus Vaccine: Fluzone® 2011-2012 Formulation
- Fluzone® High-Dose Vaccine Group (Active Comparator): Participants will receive the Influenza Virus Vaccine, Fluzone® High-Dose 2011-2012 Formulation.
  Interventions: Biological: Influenza Virus Vaccine: Fluzone® High-Dose 2011-2012 Formulation

INTERVENTIONS:
Biological: Influenza Virus Vaccine: Fluzone® 2011-2012 Formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® 2011-2012 Formulation
  Arms: Fluzone® Vaccine Group
Biological: Influenza Virus Vaccine: Fluzone® High-Dose 2011-2012 Formulation — 0.5 mL, Intramuscular
  Other Names: Fluzone® High-Dose 2011-2012 Formulation
  Arms: Fluzone® High-Dose Vaccine Group

SUMMARY:
The aim of the study is to evaluate the safety and immunogenicity of the 2011-2012 formulation of Fluzone and Fluzone High-Dose vaccines in participants aged 65 years and older.

Objectives:

* To describe the safety of Fluzone vaccine and Fluzone High-Dose vaccine among adults ≥ 65 years of age.
* To describe the immunogenicity of Fluzone vaccine and Fluzone High-Dose vaccine among adults ≥ 65 years of age.

DETAILED DESCRIPTION:
Historically, the annual safety and immunogenicity study of Fluzone vaccine has been conducted in the US in support of licenses held by sanofi pasteur in various countries.

Participants will be randomized to receive a dose of either Fluzone® or Fluzone® High-Dose vaccine and will be followed up for safety and immunogenicity. The duration of participation in the trial will be approximately 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 65 years of age on the day of inclusion.
* Informed consent form (ICF) has been signed and dated.
* Able to attend all scheduled visits and to comply with all trial procedures.

Exclusion Criteria:

* History of serious adverse reaction to any influenza vaccine.
* Receipt of any vaccine within 30 days before receiving study vaccine, or plans to receive another vaccine before the 2nd visit.
* Participation in another interventional clinical trial investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the first study vaccination or during the course of the study, unless no intervention for the other study occurred within the 30 days prior to the first study vaccination and none are planned before the subject would complete safety surveillance for the present study.
* Influenza vaccination in the 6 months preceding enrollment in the study.
* Known systemic hypersensitivity to eggs, chicken proteins, latex, or any of the vaccine components, or a history of a life-threatening reaction to Fluzone or Fluzone High-Dose vaccine or to a vaccine containing any of the same substances (the complete list of vaccine components is included in the Investigator's Brochure and/or the package insert) .
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months.
* Thrombocytopenia, which may be a contraindication for intramuscular (IM) vaccination, at the discretion of the Investigator.
* Bleeding disorder or receipt of anticoagulants in the 3 weeks preceding inclusion, which may be a contraindication for IM vaccination, at the discretion of the Investigator.
* Any condition that in the opinion of the Investigator would pose a health risk to the subject if enrolled or could interfere with the evaluation of the vaccine.
* Personal history of Guillain-Barré syndrome.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion.
* Seropositivity for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C, as reported by the subject.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Current alcohol or drug addiction that, in the opinion of the Investigator, might interfere with the ability to comply with trial procedures.
* Moderate or severe acute illness/infection (according to Investigator judgment) or febrile illness (temperature ≥ 38.0°C [≥ 100.4°F]) on the day of vaccination. A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Actual)
Dates: Start 2011-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (6):
- United States (6):
  - Colorado Springs, Colorado
  - Council Buffs, Iowa
  - Metairie, Louisiana
  - Springfield, Missouri
  - Bensalem, Pennsylvania
  - Austin, Texas

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 07 September through 24 October 2011 in 6 clinic sites in the US.
Pre-assignment Details: A total of 300 participants who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Fluzone® Vaccine Group: Participants received the Influenza Virus Vaccine: Fluzone® 2011-2012 Formulation
- Fluzone® High-Dose Vaccine Group: Participants received the Influenza Virus Vaccine, Fluzone® High-Dose 2011-2012 Formulation.
Period: Overall Study
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group
Started | 150 | 150
Completed | 150 | 150
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluzone® High-Dose Vaccine Group: Participants received the Influenza Virus Vaccine: Fluzone® High-Dose 2011-2012 Formulation.
- Total: Total of all reporting groups
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group | Total
Number analyzed (Participants) | 150 | 150 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 150 | 150 | 300
Age Continuous [Mean (Standard Deviation); unit: Months] | 72.6 (5.8) | 71.6 (4.8) | 72.1 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 92 | 183
  Male | 59 | 58 | 117
Region of Enrollment [Number; unit: Participants]
  United States | 150 | 150 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting at Least One Solicited Injection Site or Systemic Reaction Following Vaccination With One Dose of Either Fluzone® or Fluzone® High-Dose Vaccine
Description: Solicited injection site reactions: Pain, Erythema and Swelling. Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia.
  Grade 3 solicited reactions were defined as: Fever ≥ 39.0°C; Pain, Headache, Malaise and Myalgia, significant, prevents daily activities; Erythema and Swelling > 100 mm.
Time Frame: Day 0 to up to Day 28 post-vaccination
Population: Solicited injection site and systemic reactions were assessed in all enrolled and vaccinated participants, Intent-to-treat population (Safety Analysis Set).
Measure: Number; unit: Participants
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group
Number analyzed (Participants) | 150 | 150
Participants
  Any injection site Pain | 36 | 79 [0 to 0]
  Grade 3 injection site Pain | 1 | 0 [0 to 0]
  Any injection site Erythema | 7 | 13 [0 to 0]
  Grade 3 injection site Erythema | 0 | 2 [0 to 0]
  Any injection site Swelling | 4 | 10 [0 to 0]
  Grade 3 injection site Swelling | 0 | 0 [0 to 0]
  Any Fever | 2 | 1 [0 to 0]
  Grade 3 Fever | 0 | 0 [0 to 0]
  Any Headache | 26 | 25 [0 to 0]
  Grade 3 Headache | 2 | 0 [0 to 0]
  Any Malaise | 21 | 24 [0 to 0]
  Grade 3 Malaise | 5 | 0 [0 to 0]
  Any Myalgia | 25 | 44 [0 to 0]
  Grade 3 Myalgia | 3 | 1 [0 to 0]

2. Other Pre Specified Outcome: Geometric Mean Titers of Antibodies to Vaccine Antigens Before and Following Vaccination With Either Fluzone® or Fluzone® High-Dose Vaccine.
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay.
Time Frame: Day 21 post-vaccination
Population: GMTs of antibodies against Influenza vaccine antigens were determined in all enrolled and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group
Number analyzed (Participants) | 147 | 145
Titers
  A/H1N1 (Pre-vaccination; N = 147, 145) | 63.9 [50.1 to 81.5] | 57.5 [44.6 to 74.1]
  A/H1N1 (Post-vaccination; N = 147, 144) | 228 [187 to 279] | 442 [362 to 540]
  A/H3N2 (Pre-vaccination; N = 147, 145) | 104 [80.2 to 134] | 102 [78.1 to 133]
  A/H3N2 (Post-vaccination; N = 147, 145) | 384 [317 to 465] | 880 [721 to 1072]
  B (Pre-vaccination; N = 147, 145) | 32.4 [27.2 to 38.5] | 31.1 [25.8 to 37.5]
  B (Post-vaccination; N = 147, 145) | 73.0 [63.4 to 84.0] | 106 [90.2 to 125]

3. Other Pre Specified Outcome: Number of Participants With Seroconversion Following Vaccination With Either Fluzone® or Fluzone® High-Dose Vaccine
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay.
  Seroconversion was defined as either a pre-vaccination HAI titer < 1:10 and a post-vaccination titer ≥ 1:40; or a pre-vaccination titer ≥ 1:10 and a four-fold increase in post-vaccination titer.
Time Frame: Day 21 post-vaccination
Population: Seroconversion to Influenza vaccine antigens were determined in all enrolled and vaccinated participants, per-protocol population
Measure: Number; unit: Participants
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group
Number analyzed (Participants) | 147 | 145
Participants
  A/H1N1 (N = 147, 144) | 53 | 88 [0 to 0]
  A/H3N2 (N = 147, 145) | 60 | 100 [0 to 0]
  B (N = 147, 145) | 32 | 60 [0 to 0]

4. Other Pre Specified Outcome: Geometric Mean of Titer Ratios (GMTR) of Antibodies to Vaccine Antigens Before and Following Vaccination With Either Fluzone® or Fluzone® High-Dose Vaccine.
Description: Anti-influenza antibodies were measured using a hemagglutination inhibition (HAI) assay.
  Geometric mean of titer ratio is the geometric mean of the individual post-vaccination/pre-vaccination titer ratios.
Time Frame: Day 21 post-vaccination
Population: Geometric mean of titer ratios of antibodies against Influenza vaccine antigens were determined in all enrolled and vaccinated participants, per-protocol population
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group
Number analyzed (Participants) | 147 | 145
Titers
  A/H1N1 (N = 147, 144) | 3.28 [2.69 to 4.01] | 7.14 [5.61 to 9.11]
  A/H3N2 (N = 147, 145) | 3.5 [2.88 to 4.24] | 8.23 [6.45 to 10.5]
  B (N = 147, 145) | 2.13 [1.90 to 2.38] | 3.14 [2.69 to 3.67]

ADVERSE EVENTS:
Time Frame: Adverse events were recorded following vaccination (Day 0) for up to 28 days post-vaccination
Arm/Group | Fluzone® Vaccine Group | Fluzone® High-Dose Vaccine Group
Serious Adverse Events (participants affected / at risk) | 1/150 | 0/150
Other Adverse Events (participants affected / at risk) | 36/150 | 79/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® Vaccine Group (N=150) | Fluzone® High-Dose Vaccine Group (N=150)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluzone® Vaccine Group (N=150) | Fluzone® High-Dose Vaccine Group (N=150)
Injection site Pain (General disorders) | 36 (36) | 79 (79)
Injection site Erythema (General disorders) | 7 (7) | 13 (13)
Injection site Swelling (General disorders) | 4 (4) | 10 (10)
Malaise (General disorders) | 21 (21) | 24 (24)
Myalgia (Musculoskeletal and connective tissue disorders) | 25 (25) | 44 (44)
Headache (Nervous system disorders) | 26 (26) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications